CLINICAL TRIAL: NCT06651112
Title: Impacts of Psychosis and Antipsychotics on Cerebral Energy Metabolism: the ATP Project (Antipsychotic-TEP-Psychosis)
Brief Title: The ATP Project (Antipsychotic-TEP-Psychosis)
Acronym: ATP
Status: Not yet recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Collaborators: Baszucki Brain Research Fund (Other)
Responsible Party: Principal Investigator, Stephen Cunnane, Professor, Université de Sherbrooke
Other Study IDs: 2025-5589
Record Dates: First submitted 2024-10-11; First posted 2024-10-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: First Episose Psychosis; Metabolic Disease; Psychosis; Episode
Keywords: psychosis; cerebral metabolism; glucose; ketone; PET scan
MeSH Terms: conditions — Metabolic Diseases; Psychotic Disorders; Ketosis | interventions — Antipsychotic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma will be collected from whole blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- First episode psychosis: Individuals aged 18 to 35 from the Estrie region who have been evaluated by the "PEP team" (First episode psychosis intervention Team of the pschiatric department of the CIUSSS de l'Estrie-CHUS) and wish to start an antipsychotic (AP) for the treatment of a first episode of psychosis.
  Interventions: Drug: Antipsychotic drugs

INTERVENTIONS:
Drug: Antipsychotic drugs — Any Antipsychotic drugs prescripbe as standrd of care for this specific populaton

SUMMARY:
The goal of this observational study is to the early impacts of psychosis and antipsychotic medications on brain metabolism in young adults recently diagnosed with a first episode of psychosis.

The main question aims to evaluate the effect of 4 to 6 weeks of antipsychotic medication on brain metabolism measured by PET scan (cerebral uptake of 11C-Acetoacetate + 18 Fluorodeoxyglucose).

Participants will undergo a multimodal imaging protocol with other measures of psychopathology (e.g., cognition, depressive symptoms, etc.) and (metabolic marker, inflammation, etc).

ELIGIBILITY:
Inclusion Criteria:

* Admission to the PEP clinic in Estrie, either outpatient or inpatient, according to the transdiagnostic PEP model.
* Willingness to begin taking an AP (regardless of type and dose, or change in type and dose during the study).
* Ability to read and express themselves in French or English.
* Capable of understanding and signing consent.

Exclusion Criteria:

* Pregnancy, childbirth in the last 6 months, or breastfeeding.
* Presence of a metallic object in the body that is incompatible with MRI.
* Any use of APs for more than 2 continuous weeks in the past year and/or 6 weeks in a lifetime (except for aripiprazole if taken at less than 2.5 mg/day or quetiapine at less than 50 mg/day, regardless of duration or timing of the prescription).
* The following comorbidities: psychosis + borderline or intellectual disability, autism spectrum disorder, substance use disorder with decompensation, psychosis induced by a medical condition, or psychosis induced by drug use or withdrawal.
* Type 1 diabetes.
* Uncontrolled acute suicidal ideation.
* Other conditions that could interfere with participation according to the judgment of the qualified physician.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals aged 18 to 35 from the Estrie region who have been evaluated by the PEP team and wish to start an antipsychotic (AP) for the treatment of a first episode of psychosis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral metabolic rate of glucose and acetotacetate | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Cerebral metabolic rate of glucose and acetotacetate(μmol/100 g/min) quantified with PET scan with 18F-FDG tracer and 11C-AcAc
Net inflow of glucose and acetoacetate | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Net inflow of glucose and acetoacetate (k) as measured by PET scan with 18F-FDG and 11C-AcAc traceur (Kglu and Kacac, min-1)

SECONDARY OUTCOMES:
% of change in Brief Psychiatric Rating Scale | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  % of change in the Brief psychiatric Rating Scale (raw score after/raw score before*100)
Concentration of glucose | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Concentration of glucose measure in fasting plasma
Concentration of insuline | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Concentration of insulinemeasure in fasting plasma
Concentration of Hemoglobin A1C | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Concentration of HbA1C measured in fasting plasma

OTHER OUTCOMES:
Global brain volume measured by MRI | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Global brain volumes measured as global brain volumes (ml) measured by MRI
Thicknesses of the cerebral cortex | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Thicknesses of the cerebral cortex (mm) measured by MRI
Depression status measured by the score of "Calgary Depression Scale for Schizophrenia | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Score of "Calgary Depression Scale for Schizophrenia" (CDSS) . Min score 0, maximum score 27 with worsening of the patient condition with hight value
Functionning level measured by the score of the Global Assessment of functionning | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Score of the "Global Assessment of functionning (GAF). Min score 0, maximum score 100, with worsening of the patient condition with higher value
Side effet score measured by the Side Effect Rating Scale | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Score on the "Side Effect Rating Scale" UKU. Min score 0, maximum score 135 (female) 129 (male), with worsening of the side effect with higher value
Alcohol consumption measured by the score of the Alcohol Use Disorders Identification Test -AUDIT | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Alcoohol consumption as measured by the score of the Alcohol Use Disorders Identification Test AUDIT.
  Min score 0, maximum score 40, with higher alcool consumption with higher value of the score
Drug consumption measured by the score of the Drug Use Disorders Identification Test -DUDIT | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Drug consumption as measured by the score of the Drug Use Disorders Identification Test DUDIT.
  Min score 0, maximum score 40, with higher alcool consumption with higher value of the score
Average weekly hours of sport/exercise per day | BEFORE introduction of antipsychotic medicationand AFTER 4 to 6 weeks
  Average weekly hours of sport/exercise per day" as measured by question 4 of the Simple Physical Activity questionnaire SIMPAQ (hour)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cunnane, Ph.D, Principal Investigator — Université de Sherbrooke; Kevin Zemmour, MD, Principal Investigator — Université de Sherbrooke; Maggie Hahn, MD, Principal Investigator — University of Toronto
Locations (1):
- Hotel-Dieu CIUSSS de l'Estrie-CHUS, Sherbrooke, Quebec, Canada

REFERENCES:
- [Background] Cunnane SC, Trushina E, Morland C, Prigione A, Casadesus G, Andrews ZB, Beal MF, Bergersen LH, Brinton RD, de la Monte S, Eckert A, Harvey J, Jeggo R, Jhamandas JH, Kann O, la Cour CM, Martin WF, Mithieux G, Moreira PI, Murphy MP, Nave KA, Nuriel T, Oliet SHR, Saudou F, Mattson MP, Swerdlow RH, Millan MJ. Brain energy rescue: an emerging therapeutic concept for neurodegenerative disorders of ageing. Nat Rev Drug Discov. 2020 Sep;19(9):609-633. doi: 10.1038/s41573-020-0072-x. Epub 2020 Jul 24. PMID 32709961
- [Background] Croteau E, Castellano CA, Richard MA, Fortier M, Nugent S, Lepage M, Duchesne S, Whittingstall K, Turcotte EE, Bocti C, Fulop T, Cunnane SC. Ketogenic Medium Chain Triglycerides Increase Brain Energy Metabolism in Alzheimer's Disease. J Alzheimers Dis. 2018;64(2):551-561. doi: 10.3233/JAD-180202. PMID 29914035
- [Background] Croteau E, Castellano CA, Fortier M, Bocti C, Fulop T, Paquet N, Cunnane SC. A cross-sectional comparison of brain glucose and ketone metabolism in cognitively healthy older adults, mild cognitive impairment and early Alzheimer's disease. Exp Gerontol. 2018 Jul 1;107:18-26. doi: 10.1016/j.exger.2017.07.004. Epub 2017 Jul 12. PMID 28709938
- [Background] Agarwal SM, Kowalchuk C, Castellani L, Costa-Dookhan KA, Caravaggio F, Asgariroozbehani R, Chintoh A, Graff-Guerrero A, Hahn M. Brain insulin action: Implications for the treatment of schizophrenia. Neuropharmacology. 2020 May 15;168:107655. doi: 10.1016/j.neuropharm.2019.05.032. Epub 2019 May 29. PMID 31152767
- [Background] Fortier M, Castellano CA, St-Pierre V, Myette-Cote E, Langlois F, Roy M, Morin MC, Bocti C, Fulop T, Godin JP, Delannoy C, Cuenoud B, Cunnane SC. A ketogenic drink improves cognition in mild cognitive impairment: Results of a 6-month RCT. Alzheimers Dement. 2021 Mar;17(3):543-552. doi: 10.1002/alz.12206. Epub 2020 Oct 26. PMID 33103819
- [Background] Andreasen NC, O'Leary DS, Flaum M, Nopoulos P, Watkins GL, Boles Ponto LL, Hichwa RD. Hypofrontality in schizophrenia: distributed dysfunctional circuits in neuroleptic-naive patients. Lancet. 1997 Jun 14;349(9067):1730-4. doi: 10.1016/s0140-6736(96)08258-x. PMID 9193383
- [Background] Townsend L, Pillinger T, Selvaggi P, Veronese M, Turkheimer F, Howes O. Brain glucose metabolism in schizophrenia: a systematic review and meta-analysis of 18FDG-PET studies in schizophrenia. Psychol Med. 2023 Aug;53(11):4880-4897. doi: 10.1017/S003329172200174X. Epub 2022 Jun 22. PMID 35730361
- [Background] Henkel ND, Wu X, O'Donovan SM, Devine EA, Jiron JM, Rowland LM, Sarnyai Z, Ramsey AJ, Wen Z, Hahn MK, McCullumsmith RE. Schizophrenia: a disorder of broken brain bioenergetics. Mol Psychiatry. 2022 May;27(5):2393-2404. doi: 10.1038/s41380-022-01494-x. Epub 2022 Mar 9. PMID 35264726
- [Background] Lee J, Xue X, Au E, McIntyre WB, Asgariroozbehani R, Panganiban K, Tseng GC, Papoulias M, Smith E, Monteiro J, Shah D, Maksyutynska K, Cavalier S, Radoncic E, Prasad F, Agarwal SM, Mccullumsmith R, Freyberg Z, Logan RW, Hahn MK. Glucose dysregulation in antipsychotic-naive first-episode psychosis: in silico exploration of gene expression signatures. Transl Psychiatry. 2024 Jan 10;14(1):19. doi: 10.1038/s41398-023-02716-8. PMID 38199991
- [Background] Agarwal SM, Stogios N, Ahsan ZA, Lockwood JT, Duncan MJ, Takeuchi H, Cohn T, Taylor VH, Remington G, Faulkner GEJ, Hahn M. Pharmacological interventions for prevention of weight gain in people with schizophrenia. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013337. doi: 10.1002/14651858.CD013337.pub2. PMID 36190739
- [Background] Raben AT, Marshe VS, Chintoh A, Gorbovskaya I, Muller DJ, Hahn MK. The Complex Relationship between Antipsychotic-Induced Weight Gain and Therapeutic Benefits: A Systematic Review and Implications for Treatment. Front Neurosci. 2018 Jan 22;11:741. doi: 10.3389/fnins.2017.00741. eCollection 2017. PMID 29403343
- [Background] Vancampfort D, Stubbs B, Mitchell AJ, De Hert M, Wampers M, Ward PB, Rosenbaum S, Correll CU. Risk of metabolic syndrome and its components in people with schizophrenia and related psychotic disorders, bipolar disorder and major depressive disorder: a systematic review and meta-analysis. World Psychiatry. 2015 Oct;14(3):339-47. doi: 10.1002/wps.20252. PMID 26407790
- [Background] Sabe M, Pallis K, Solmi M, Crippa A, Sentissi O, Kaiser S. Comparative Effects of 11 Antipsychotics on Weight Gain and Metabolic Function in Patients With Acute Schizophrenia: A Dose-Response Meta-Analysis. J Clin Psychiatry. 2023 Feb 8;84(2):22r14490. doi: 10.4088/JCP.22r14490. PMID 36752753
- [Background] Fan Z, Wu Y, Shen J, Ji T, Zhan R. Schizophrenia and the risk of cardiovascular diseases: a meta-analysis of thirteen cohort studies. J Psychiatr Res. 2013 Nov;47(11):1549-56. doi: 10.1016/j.jpsychires.2013.07.011. Epub 2013 Aug 15. PMID 23953755
- [Background] Correll CU, Hojlund M, Graham C, Todtenkopf MS, McDonnell D, Simmons A. Weight Gain and Metabolic Changes in Patients With First-Episode Psychosis or Early-Phase Schizophrenia Treated With Olanzapine: A Meta-Analysis. Int J Neuropsychopharmacol. 2023 Jul 31;26(7):451-464. doi: 10.1093/ijnp/pyad029. PMID 37326421